CLINICAL TRIAL: NCT06005493
Title: A Phase I/II Open-label Dose Escalation and Dose Expansion Study to Evaluate the Safety, Pharmacokinetics, Pharmacodynamics, and Efficacy of AZD5863, a T Cell-engaging Bispecific Antibody That Targets Claudin 18.2 (CLDN18.2) and CD3 in Adult Participants With Advanced or Metastatic Solid Tumors
Brief Title: Study of AZD5863 in Adult Participants With Advanced or Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: D9750C00001; 2023-504139-42-00 (Registry Identifier: CTIS); 2023-000154-20 (EudraCT Number)
Record Dates: First submitted 2023-06-16; First posted 2023-08-22 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-11

CONDITIONS: Gastric Cancer; Gastro-esophageal Junction Cancer; Pancreatic Ductal Adenocarcinoma; Esophageal Adenocarcinoma
Keywords: CLDN18.2 / Claudin 18.2; CD3; T cell-engaging bi-specific antibody; Gastric cancer; Gastro-esophageal junction cancer; Pancreatic ductal adenocarcinoma; Solid tumors; AZD5863
MeSH Terms: conditions — Stomach Neoplasms; Adenocarcinoma Of Esophagus

STUDY DESIGN:
Intervention Model Description: The study consists of individual modules each evaluating the safety and tolerability of AZD5863 dosed as monotherapy:
  * Module 1: AZD5863 intravenous administration
  * Module 2: AZD5863 subcutaneous administration
  Modules 1 and 2 each consist of two parts: Part A, Dose Escalation and Part B, Dose Expansion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Module 1: AZD5863 Monotherapy Intravenous (IV) (Experimental): Module 1: AZD5863 Intravenous (IV) Monotherapy
  Interventions: Drug: AZD5863
- Module 2: AZD5863 Monotherapy Subcutaneous (SC) (Experimental): Module 2: AZD5863 Subcutaneous (SC) Monotherapy
  Interventions: Drug: AZD5863

INTERVENTIONS:
Drug: AZD5863 — T cell-engaging bi-specific antibody that targets CLDN18.2 (Claudin18.2) on tumor cells and CD3 on T cells

SUMMARY:
This research is designed to determine if experimental treatment with AZD5863, a T cell-engaging bispecific antibody that targets Claudin 18.2 (CLDN18.2) and CD3, is safe, tolerable and has anti-cancer activity in patients with advanced solid tumors.

DETAILED DESCRIPTION:
This is a first-time in human, modular Phase I/II, open-label multicentre study of AZD5863 monotherapy administered intravenously (Module 1), or AZD5863 monotherapy administered subcutaneously (Module 2) in patients with advanced or metastatic solid tumors. Each module contains dose-escalation (Part A) and dose-expansion (Part B).

ELIGIBILITY:
Key Inclusion Criteria:

* Age ≥ 18 at the time of signing the informed consent
* Histologically confirmed diagnosis of adenocarcinoma of the stomach, gastro-esophageal junction, esophagus, or pancreas
* Must have at least one measurable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
* Must show positive CLDN18.2 expression in tumor cells as determined by central immunohistochemistry (IHC)
* Eastern Cooperative Oncology Group Performance status (ECOG PS): 0-1 at screening
* Predicted life expectancy of ≥ 12 weeks
* Adequate organ and bone marrow function measured within 28 days prior to first dose as defined by the protocol
* Contraceptive use by men or women should be consistent with local regulations, as defined by the protocol
* Must have received at least one prior line of systemic therapy in the advanced/metastatic setting

Key Exclusion Criteria:

* Unresolved toxicity from prior anticancer therapy of Common Terminology Criteria for Adverse Events (CTCAE) Grade ≥ 2 except for those defined by the protocol
* Participant experienced unacceptable cytokine release syndrome (CRS) or Immune Effector Cell Associated Neurotoxicity (ICANS) following prior T cell engagers (TCE) or chimeric antigen receptor T (CAR-T) cell therapy
* Previous history of hemophagocytic lymphohistiocytosis (HLH) / macrophage activation syndrome (MAS)
* Active or prior documented autoimmune or inflammatory disorders within 3 years of start of treatment
* central nervous system (CNS) metastases or CNS pathology, as defined by the protocol, within 3 months prior to consent
* Infectious disease including active human immunodeficiency virus (HIV), active hepatitis B/C, uncontrolled infection with EBV, uncontrolled active systemic fungal, bacterial or other infection
* Cardiac conditions as defined by the protocol
* History of thromboembolic event within the past 3 months prior to the scheduled first dose of study intervention
* Participant requires chronic immunosuppressive therapy
* Participants on anticoagulation therapy with long-acting anticoagulants or other class of anticoagulants at therapeutic doses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2023-07-11 (Actual); Primary Completion 2027-07-16 (Estimated); Study Completion 2027-07-16 (Estimated)

PRIMARY OUTCOMES:
The number of patients with adverse events | From first dose of study drug up to 90 days post last dose and prior to start of subsequent anticancer therapy
  Number of patients with adverse events by system organ class and preferred term
The number of patients with adverse events of special interest | From first dose of study drug up to 90 days post last dose and prior to start of subsequent anticancer therapy
  Number of patients with adverse events of special interest by system organ class and preferred term
The number of patients with dose-limiting toxicity (DLT), as defined in the protocol. | From first dose of study drug until the end of Cycle 1
  A DLT is a toxicity as defined in the protocol that occurs from the first dose of study drug up to and including the planned end of Cycle 1 (the DLT assessment period) that is assessed as unrelated to the disease or disease-related processes under investigation.
The number of patients with serious adverse events | From first dose of study drug up to 90 days post last dose and prior to start of subsequent anticancer therapy
  Number of patients with serious adverse events by system organ class and preferred term
Objective Response Rate (ORR) | From first dose of study drug to progressive disease or death in the absence of disease progression (approx. 2 years)
  The percentage of patients with a confirmed investigator assessed complete or partial response according to response criteria in solid tumours (RECIST 1.1). Dose expansion only.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | From first dose of study drug to progressive disease or death in the absence of disease progression (approx. 2 years)
  The percentage of patients with a confirmed investigator assessed complete or partial response according to response criteria in solid tumours (RECIST 1.1). Dose escalation only.
Disease Control Rate (DCR) | From first dose of study drug to progressive disease or death in the absence of disease progression (approx. 2 years)
  Percentage of patients with confirmed complete or partial response or having stable disease maintained for >= 11 weeks from first dose, according to response criteria in solid tumours (RECIST 1.1).
Duration of response (DoR) | From the first documented response to progressive disease or death in the absence of disease progression (approx. 2 years)
  The time from the date of first response until date of disease progression or death in the absence of disease progression, according to response criteria in solid tumours (RECIST 1.1).
Progression free Survival (PFS) | From the start of study treatment/date of randomization to progressive disease or death in the absence of disease progression (approx. 2 years)
  The time from the start of study treatment/date of randomization until RECIST 1.1 defined disease progression or death in the absence of disease progression.
Overall Survival (OS) | From the start of study treatment/date of randomization to death (to be followed-up for approx. 2 years)
  The time from the start of study treatment/date of randomization until death due to any cause.
Pharmacokinetics of AZD5863: Maximum plasma concentration of the study drug (Cmax) | From the first dose of study intervention, at predefined intervals throughout the study (approx. 2 years)
  Maximum observed plasma concentration of the study drug
Pharmacokinetics of AZD5863: Area Under the concentration-time curve (AUC) | From the first dose of study intervention, at predefined intervals throughout the study (approx. 2 years)
  Area under the plasma concentration-time curve
Pharmacokinetics of AZD5863: Clearance | From the first dose of study intervention, at predefined intervals throughout the study (approx. 2 years)
  A pharmacokinetic measurement of the volume of plasma from which the study drug is completely removed per unit time.
Pharmacokinetics of AZD5863: Terminal elimination half-life (t 1/2) | From the first dose of study intervention, at predefined intervals throughout the study (approx. 2 years)
  Terminal elimination half life.
Immunogenicity of AZD5863 | From the first dose of study intervention, at predefined intervals throughout the study (approx. 2 years)
  The number and percentage of participants who develop anti-drug antibodies (ADAs) measured in serum
Preliminary antitumor activity with target expression pre- and post-delivery of AZD5863 | From time of Informed consent, at predefined intervals (including screening, on-treatment or end of treatment) throughout the study (over approx. 2 years)
  Measure CLDN18.2 expression (IHC) in baseline and/or on-treatment tumor biopsies and correlate with clinical outcome

CONTACTS AND LOCATIONS:
Locations (21):
- United States (3):
  - Research Site, Jacksonville, Florida
  - Research Site, Rochester, Minnesota
  - Research Site, New York, New York
- China (2):
  - Research Site, Beijing
  - Research Site, Shandong
- France (2):
  - Research Site, Toulouse
  - Research Site, Villejuif
- Japan (3):
  - Research Site, Chūōku
  - Research Site, Kashiwa
  - Research Site, Kōtoku
- Netherlands (3):
  - Research Site, Amsterdam
  - Research Site, Groningen
  - Research Site, Rotterdam
- Research Site, Seoul, South Korea
- Taiwan (3):
  - Research Site, Kaohsiung City
  - Research Site, Tainan
  - Research Site, Taoyuan District
- United Kingdom (4):
  - Research Site, Dundee
  - Research Site, London
  - Research Site, Metropolitan Borough of Wirral
  - Research Site, Oxford

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
  "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Gaspar M, Natoli M, Castan L, Rahmy S, Korade M 3rd, Kelton C, Mulgrew K, Huhn O, Rees DG, Sigurdardottir A, Lloyd C, Taylor JJ, Brailey PM, Dallaway L, Toloczko A, Giraldo N, Broggi MAS, Kunihiro A, Abhishek S, He Y, Rong Y, Eyles J, Ball K, Fitzgerald J, Hammond SA, Cemerski S, Dovedi SJ, Cobbold M. An affinity-modulated T cell engager targeting Claudin 18.2 shows potent anti-tumor activity with limited cytokine release. J Immunother Cancer. 2025 Aug 4;13(8):e011857. doi: 10.1136/jitc-2025-011857. PMID 40759445